CLINICAL TRIAL: NCT06424860
Title: Dietary Fish Oil and Metformin Intervention for Heart Health in PCOS
Brief Title: Fish Oil, Metformin and Heart Health in PCOS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00141704
Record Dates: First submitted 2024-04-29; First posted 2024-05-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: PCOS; Cardiovascular Disease; Atherosclerotic Cardiovascular Disease; Atherosclerotic Plaque; Cardiac Hypertrophy
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Plaque, Atherosclerotic; Cardiomegaly | interventions — Fish Oils; Metformin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Active Comparator): metformin (1500mg/d) and placebo (olive oil capsule)
  Interventions: Drug: Metformin
- Fishoil and metformin (Experimental): metformin (1500mg/d) and fish oil (4000mg/d)
  Interventions: Dietary Supplement: Fish oil; Combination Product: Fish Oil and Metformin

INTERVENTIONS:
Dietary Supplement: Fish oil — For 12 months
  Arms: Fishoil and metformin
Drug: Metformin — 12 months
  Arms: Metformin
Combination Product: Fish Oil and Metformin — 12 months
  Arms: Fishoil and metformin

SUMMARY:
Women with Polycystic Ovary Syndrome (PCOS) have high testosterone levels which is associated with altered insulin-glucose metabolism and an adverse blood lipid profile, predisposing them to the development of Type II Diabetes and Cardiovascular Disease (CVD). This study will investigate the use of dietary fish oil supplementation as a safe and effective intervention, and as an adjunct therapy to standard of care treatment with metformin to improve heart health, blood lipids and insulin-glucose metabolism in women with PCOS, and those with PCOS and Type 2 Diabetes.

DETAILED DESCRIPTION:
OBJECTIVES The objective in this proposed study is to determine the effect of dietary fish oil supplementation with metformin compared to standard of care metformin-alone treatment for 12 months on plasma lipids and apoB- remnant lipoprotein metabolism, and atherosclerotic cardiovascular disease and cardiac function in high-risk overweight-obese young individuals with PCOS.

This study will provide evidence-based research on the efficacy of fish oil, in the form as an adjunct therapy to standard treatment with metformin, as a safe nutritional treatment to add to therapeutic guidelines to reduce early CVD risk in young women with PCOS.

Specific Objectives;

1. To quantify carotid intimal medical thickness (cIMT) and plaque height before and after the intervention to assess the effect of fish oil supplementation combined with metformin standard of care on atherosclerotic cardiovascular disease and cardiac function.
2. To determine the effects of dietary fish oil supplementation combined with metformin and metformin standard of care on fasting and non-fasting plasma TG, apoB48 and apoB100-lipoprotein concentrations, and cardiac function variables including left ventricular (LV) posterior wall thickness, LV ejection fraction.
3. To assess the effect of dietary fish oil supplementation on insulin, glucose, and endocrine parameters.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PCOS
* overweight-obese (BMI >25 kg/m2)
* elevated fasting plasma TG (>150 mg/dL)
* and/or apoB48-remnant cholesterol lipoproteins (>20 ug/ml)
* impaired insulin sensitivity (glucose 100-125 mg/dL and/or insulin >15 (uM/ml), and may be diagnosed with T2D (blood glucose >126 mg/dL).

Exclusion Criteria:

-pregnancy, lactation

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Carotid intimal medial thickness | 12 months
  mm
carotid plaque height | 12 months
  mm
Left ventricular global longitudinal strain (LVGLS) | 12 months
  percent change in LVGLS

SECONDARY OUTCOMES:
Blood lipids | 12 months
  TG, LDL-C, HDL-C, non-HDL-C mmol/l
ApoB-lipoproteins | 12 months
  apob48 and apoB100 mg/l
remnant-cholesterol | 12 months
  mmol/l
Testosterone | 12 months
  nmol/l
insulin | 12 months
  pmol/l
glucose | 12 months
  mmol/l

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Human Nutrition Research Unit - Li Ka Shing Health Research Center, Edmonton, Alberta
  - Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - University of Alberta Hospital - Division of Endocrinology, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No
no plan